CLINICAL TRIAL: NCT04280913
Title: Clinical Outcomes of Hospitalized Patients With Coronavirus Disease 2019
Brief Title: Clinical Outcomes of Patients With COVID19
Status: Withdrawn | Type: Observational
Why Stopped: The research project was changed.
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Huizhou Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, LuQian Zhou, Principal Investigator, Guangzhou Institute of Respiratory Disease
Other Study IDs: GZHZ-COVID19
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Hospitalized patients with COVID-19
  Interventions: Other: retrospective analysis

INTERVENTIONS:
Other: retrospective analysis — The investigators retrospectively analyzed the hospitalized patients with COVID-19.

SUMMARY:
As of February 17th, 2020, China has 70635 confirmed cases of coronavirus disease 2019 (COVID-19), including 1772 deaths. Human-to-human spread of virus via respiratory droplets is currently considered to be the main route of transmission. The number of patients increased rapidly but the impact factors of clinical outcomes among hospitalized patients are still unclear.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with COVID19

Exclusion Criteria:

* Suspected patients with COVID19, not confirmed by the laboratory
* Patients who are refused to receive medical treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective study of hospitalized patients with COVID19.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to negative conversion of severe acute respiratory syndrome coronavirus 2 | 1 month
  The primary outcome is the time to negative conversion of coronavirus

SECONDARY OUTCOMES:
Length of stay in hospital | 1 month
  The time of hospitalization.
Survival | 1 month
  The rate of survival within hospitalization of these patients will be tracked.
Intubation | 1 month
  The rate of intubation within hospitalization of these patients will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Luqian Zhou, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- HuiZhou Municipal Central Hospital, Huizhou, Guangdong, China